CLINICAL TRIAL: NCT00970125
Title: Using Video Images to Improve Advance Care Planning in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, Faculty, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008-P-002156/2; R21CA139121-01 (NIH)
Record Dates: First submitted 2009-08-06; First posted 2009-09-02 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Advanced Cancer
Keywords: advance care planning; cancer
MeSH Terms: conditions — Neoplasms | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cancer subjects (Experimental)
  Interventions: Behavioral: video

INTERVENTIONS:
Behavioral: video — outline of the goals of care

SUMMARY:
The purpose of this study is to study whether preferences for the goals of care for 80 subjects with end-stage cancer are altered after viewing a video outlining the goals of care compared to their initial preferences after hearing a verbal description of the goals of care alone.

DETAILED DESCRIPTION:
The purpose of this study is to study whether preferences for the goals of care for 80 subjects with end-stage cancer are altered after viewing a video outlining the goals of care compared to their initial preferences after hearing a verbal description of the goals of care alone. Subjects will choose among three goals of care, life prolonging care, basic medical care, and comfort care.

ELIGIBILITY:
Inclusion Criteria:

1. Terminal, progressive cancer with poor prognosis whose treatment intent is palliative, based on the following definition:

   * All patients with brain cancer, liver cancer, inoperable non-small cell lung carcinoma, pancreatic cancer, or gallbladder cancer; OR
   * Patients with the following cancers: metastatic colon cancer or stage III or IV non-small cell lung cancer; OR
   * Patients with the following cancers, if first-line therapy has failed and limited response is expected to second-line therapy: breast cancer, colorectal cancer, head and neck cancer, stomach cancer, esophageal cancer, melanoma, leukemia, ovarian cancer, prostate cancer, renal cancer, sarcoma, lung cancer, myeloma, or lymphoma.
   * The terms terminal, progressive, poor prognosis, palliative intent and limited response will be judged by the patient's oncologist (and not by the RSA or consenting professional).
2. Return patient visit (defined as a patient known to the oncologist from previous assessments and treatments, where the working and personal relationship has been established and not a new patient to the clinic).
3. English speaking. Only English-speaking patients will be included in our present study since English is the validated language of our study tools.
4. Given the sensitive nature of the study, clinicians will decide whether the patient is a potentially appropriate subject based on their knowledge of the patient.
5. Able to provide informed consent.
6. Age greater than or equal to 21.

Exclusion Criteria:

1. MMSE < 25.
2. Psychological state not appropriate for end-of-life discussion as determined by the treating clinician.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
end of life preference at time of interview | 5 minutes after survey

SECONDARY OUTCOMES:
knowledge | 5 minutes after survey
decisional conflict | 5 minutes after survey

CONTACTS AND LOCATIONS:
Overall Officials: Angelo E. Volandes, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Memorial Sloan Kettering, New York, New York, United States